CLINICAL TRIAL: NCT00018694
Title: Biologic Significance of Cholestanol in Man
Brief Title: Cholestanol in Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None
Other Study IDs: GAST-007-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Cerebrotendinous Xanthomatosis
Keywords: bile acid synthesis; chenodeoxycholic acid; sterol 27-hydroxylase
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous | interventions — Chenodeoxycholic Acid

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Chenodeoxycholic Acid

INTERVENTIONS:
Drug: Chenodeoxycholic Acid

SUMMARY:
The treatment of cerebrotendinous xanthomatosis an in born error of bile acid synthesis with chenodeoxycholic acid. Patients with this disease over produce cholestanol and bile acid precursors because of the block in synthesis. Replacement with chenodeoxycholic acid shut down abnormal pathway and reduces elevated level of cholestanol and improves the clinical syndrome.

DETAILED DESCRIPTION:
Cerebrotendinous xanthomatosis is a recessively inherited in born of bile acid synthesis due to a mutation in sterol 27-hydroxylase (CYP27A1). Patients with this disease suffer from xanthomas located in the brain and tendon, accelerated atherosclerosis progression neurologic disease and cataracts. Plasma cholesterol levels are normal but cholestanol and C-27 bile alcohol that precursor of bile acid synthesis accumulate and are believe are responsible for the atherosclerosis, xanthomas and neurologic disease. Analysis of the bile reveal a severe sufficiency of the primary bile acid chenodeoxycholic acid that can not be produce because of the inherited defect. However, replacement of chenodeoxycholic acid in the enterohepatic pool inhibit abnormal bile acid synthesis and reduces the elevated level of cholestanol and C-27 bile alcohol this therapy halt the neurologic disease and prevents symptomatic atherosclerosis developing.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical and biochemical findings of cerebrotendinous xanthomatosis. Elevated levels of serum cholestanol and bile acid precursors.

Exclusion Criteria:

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Salen, Principal Investigator — VA New Jersey Health Care System, East Orange
Locations (1):
- VA New Jersey Health Care System, East Orange, East Orange, New Jersey, United States